CLINICAL TRIAL: NCT03523195
Title: Physical Activity After Cancer Treatment (PACT): Pilot Study of Exercise in Stage II-III Breast Cancer Survivors
Brief Title: Exercise Intervention After Cancer Treatment for Improving Health in Stage II-III Breast Cancer Survivors
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 9988; NCI-2018-00544 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9988 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Cancer Survivor; Estrogen Receptor Positive; HER2/Neu Negative; Progesterone Receptor Positive; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Monitoring, Physiologic; Exercise Test

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 0 (written information) (Active Comparator): Participants wear Fitbit and receive written information on healthy exercise and diet recommendations.
  Interventions: Other: Informational Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Questionnaire Administration; Other: Physical Performance Testing
- Arm I (exercise program) (Experimental): Participants complete exercise program including aerobic and resistance exercises over 60 minutes 3 times per week for 12 weeks. Exercise is supervised all 3 times during weeks 1-2. During weeks 3-12, exercise is supervised 2 times a week, with home-based coaching for an additional 60 minutes a week.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Other: Physical Performance Testing

INTERVENTIONS:
Behavioral: Exercise Intervention — Complete exercise program
  Arms: Arm I (exercise program)
Other: Informational Intervention — Receive written information on healthy exercise and diet recommendations
  Arms: Arm 0 (written information)
Other: Laboratory Biomarker Analysis — Blood tests
Device: Monitoring Device — Wear Fitbit
  Other Names: Monitor
  Arms: Arm 0 (written information)
Other: Questionnaire Administration — Ancillary studies
Other: Physical Performance Testing — Performance of physical tests
  Other Names: Physical Function Testing

SUMMARY:
This pilot trial studies how well exercise intervention after cancer treatment works in improving physical activity in stage II-III breast cancer survivors. An exercise intervention may promote regular physical activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the adherence rate of the experimental exercise program, and deem as feasible if at least 80% of participants complete 80% or more of a 12-week, 180 minute aerobic+resistance training program that combines structured, individualized onsite exercise at the Fred Hutch Prevention Center with at-home exercise.

II. Identify up to 5 circulating micro ribonucleic acid (c-miRNA) biomarkers that show the largest differential change from baseline when comparing levels in the exercise program to those in the Fitbit-activity control condition.

SECONDARY OBJECTIVES:

I. Explore associations between changes in miRNAs and serum biomarkers (IL-6, lipids, adiponectin and leptin, C-reactive protein [CRP]) and physiological outcomes (resting heart rate, blood pressure, 1 repetition max, 6 minute walk, timed up and go test) of the exercise program.

II. Explore changes in the patient-reported outcomes (PRO) in response to the exercise intervention relative to the control group, and finalize measures to use in the design of the phase III clinical trial based on descriptive changes from baseline to follow-ups in the intervention versus (vs.) control groups.

OUTLINE: Participants are randomized into 1 of 2 arms.

ARM 0: Participants wear Fitbit and receive written information on healthy exercise and diet recommendations.

ARM 1: Participants complete exercise program including aerobic and resistance exercises over 60 minutes 3 times per week for 12 weeks. Exercise is supervised all 3 times during weeks 1-2. During weeks 3-12, exercise is supervised 2 times a week, with home-based coaching for an additional 60 minutes a week.

ELIGIBILITY:
Inclusion Criteria:

* Single malignancy with diagnosis of breast cancer diagnosis of stage II-III, estrogen and progesterone positive, HER-2neu negative, and on stable dose of aromatase inhibitor (AI) for past 3 months, with AI expected to be stable for the study duration
* No evidence of disease
* 1-5 years post active treatment for malignancy
* Body mass index 19 to 35
* Sedentary (< 100 minutes of moderate intensity exercise per week)
* English adequate to complete assessments and follow exercise instructions
* Able to independently use transportation to attend 2-day a week onsite exercise training
* Access to a computer or smartphone

Exclusion Criteria:

* Current tobacco use or electronic cigarette smoker
* Pregnant
* Diabetes requiring insulin injection
* Lymphedema that restricts range of motion or with worsening symptoms in the past month, or without compression garment
* Weight change of more than 10 pounds in previous 3 months will exclude from study participation at baseline
* Medical or other issue impacting exercise ability or safety, or ability to comply with study procedures (e.g. significant vision or cognitive impairment, major illness, in hospital or other institution), and specifically:

  * Have been hospitalized within 3 months prior to screening for major atherosclerotic events (e.g. myocardial infarction, target-vessel revascularization, coronary bypass surgery, stroke or blood clot) or other major medical condition (as determined by an investigator) that may put the subject at risk because of his/her participation in the study;
  * Have an implanted cardiac pacemaker or other implanted cardiac device;
  * Have chronic, uncontrolled hypertension as judged by the investigator;
  * Have a creatinine clearance < 45 mL/min as calculated by the Cockcroft-Gault equation;
  * Subject's hand or legs have mobility impairment from fractures, arthritis, surgery, muscle disease or other injury that may interfere with any study procedure or ability to exercise

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Adherence | Up to 26 weeks
  Will assess the percent of expected onsite sessions attended by participants as determined by Prevention Center attendance log.
Differential micro ribonucleic acid expression | At baseline, 13, and 26 weeks
  Will compare between arms. Descriptive statistics will be provided. Will calculate the log-fold change between baseline measure and post-baseline measure, and the difference in the log-fold change will be calculated between the two arms.

SECONDARY OUTCOMES:
Percent of expected home exercise sessions completed as determined by the home exercise logs for those choosing to not come in for a third weekly session | Up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Syrjala, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Julie Gralow, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Marie-Laure Crouch, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States